CLINICAL TRIAL: NCT00507910
Title: Pes Planus After Weber B and C Ankle Fractures
Brief Title: The Development of Flat Foot After Ankle Fractures
Status: Completed | Type: Observational
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Dr. Allan Giachino, MD, Ottawa Hospital Research Institute
Other Study IDs: OHREB2006542
Record Dates: First submitted 2007-07-25; First posted 2007-07-27 (Estimated); Last update posted 2011-07-21 (Estimated); Status verified 2011-07

CONDITIONS: Pes Planus
Keywords: ankle fracture; pes planus
MeSH Terms: conditions — Flatfoot; Ankle Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
In this study we are trying to determine the incidence of flat foot (also called pes planus) among patients who have had an ankle fracture. As compared to the general population, it is predicted that the incidence of pes planus will be higher among people who have fractured their ankle.

DETAILED DESCRIPTION:
Pes planus may develop following ankle fractures due to additional injuries that are sustained at the time of ankle fracture. If this study can demonstrate an association, further research would investigate how to effectively treat the pes planus early to prevent it from becoming a symptomatic problem.

ELIGIBILITY:
Inclusion Criteria:

Patients will be considered eligible if:

* They have sustained Weber type B or C ankle fractures and needed open reduction
* They are 18 years of age or older
* They are expected to be full weight bearing for at least 4 months to allow the potential of supporting structures to stretch and pes planus to develop

Exclusion Criteria:

* Patients will be excluded if they already have flat foot in their non-fractured foot.
* Patients with bilateral ankle fractures
* Patients who are not competent to sign a consent form
* A second fracture to the ankle
* Pathological fractures
* Patients with underlying cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2006-12; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alan Giachino, Principal Investigator — OHRI
Locations (1):
- The Ottawa Hospital, Ottawa, Ontario, Canada